CLINICAL TRIAL: NCT01146782
Title: The ATLAST Trial - A Multicenter, Prospective Study of the Attune Sleep Apnea System for the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: Study of a Sleep Apnea System for the Treatment of Obstructive Sleep Apnea
Acronym: ATLAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ApniCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 10753
Record Dates: First submitted 2010-06-15; First posted 2010-06-22 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Treatment with the Attune Sleep Apnea System
  Interventions: Device: Attune Sleep Apnea System

INTERVENTIONS:
Device: Attune Sleep Apnea System — Console and mouthpiece sleep apnea system

SUMMARY:
This is a prospective study of the Attune Sleep Apnea System for the treatment of obstructive sleep apnea. The objective of the study is to demonstrate safety and effectiveness of the Attune Sleep Apnea System to support FDA marketing clearance of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages of 18 and 80.
2. Diagnosis of OSA, based on ODI 10-60 (as assessed per home screening night).
3. Subject is fluent in English and understands the Study protocol and is willing and able to comply with Study requirements and sign the informed consent form.
4. BMI < 40.
5. Subject has a least one molar in each of the four quadrants of the mouth (right upper, right lower, left upper, and left lower).
6. Subject has proper mouthpiece fit, as assessed by home screening night (See section 8.3).

Exclusion Criteria:

1. OSA treatment within two weeks prior to Medical/Dental screening visit.
2. Poor nasal patency as evidenced by Peak Nasal Inspiratory Flow (PNIF) less than 75 l/min (assessed at baseline medical visit). In addition, any ongoing process or condition that limits nasal breathing or indications thereof, including: obligate mouth-breathing, persistent blockage of one or both nostrils resulting in the inability to sleep with the mouth closed, chronic nasal congestion, chronic allergic rhinitis, and intermittent allergic rhinitis that does not respond to non-sedating/non-stimulating medical therapy.
3. Oral cavity infection or any other oral or dental condition or problem that would limit subject use of the Attune Sleep Apnea System (e.g. dentures, loose tooth/teeth, temporomandibular joint (TMJ) conditions, or any oral or dental condition that the Investigator believes could be exacerbated by the Attune Sleep Apnea System.
4. Prior use of the Attune Sleep Apnea System.
5. History of any OSA surgical treatment including uvulopalatopharyngoplasty surgery (UPPP), maxillomandibular advancement surgery (MMA), radio frequency (RF) ablation treatment, palatal stent devices, etc.
6. Current use or use within the previous 2 weeks of medications or other agents that may affect sleep or PSG, including:

   1. Hypnotics, anxiolytics, anticonvulsants, sedating antihistamines, stimulants, sedating antidepressants or other medications likely to affect neurocognitive function and/or alertness. Patients on stable selective serotonin reuptake inhibitor (SSRI) therapy for > 3 months and who are expected to remain on therapy for the Study duration, may continue SSRI treatment.
   2. Consumption of > 500mg caffeine per day (e.g. > 8 cola-type beverages, > 5 cups of coffee).
   3. Any known illicit drug use or abuse within the past year, or failure to pass drug urine screen test, or alcohol breathalyzer test with result over 0.05% BAL.
   4. Smokers who smoke during the night (interference with PSG).
7. Any concomitant diagnosed or suspected sleep or chronic neurological disorders, other than OSA, including insomnia, and central sleep apnea.
8. Currently working nights, rotating night shifts, planned travel across four or more time zones required during Study period, or within two weeks prior to Study enrollment, or sleep schedule not compatible with sleep lab practices.
9. Potential sleep apnea complications that, in the opinion of the investigator, may affect the health or safety of the participant, including: low blood oxygen, recent near-miss or prior automobile accident due to sleepiness, reported history of severe cardiovascular disease (including NYHA class III or IV heart failure, CAD with angina or MI/stroke in past 6 months, uncontrolled hypertension or hypotension, cardiac arrhythmias), reported respiratory disorders, or use of medication or other treatment which may pose additional risk to the subject or confound the results of the Study.
10. Female subjects who are pregnant or intend to become pregnant during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Colrain, PhD, Principal Investigator — Stanford Reasearch Institute (SRI)
Locations (6):
- United States (6):
  - REM Medical, Phoenix, Arizona
  - Peninsula Sleep Center, Burlingame, California
  - SRI, Menlo Park, California
  - Sleep Disorders Center of Georgia (SDCG), Atlanta, Georgia
  - SleepMed, Columbia, South Carolina
  - Sleep Medicine Associates of Texas (SMAT), Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects for the study were recruited from the Investigator's sleep clinic or through advertising. Advertisements were approved by the applicable Institutional Review Board (IRB) prior to use.
Pre-assignment Details: Initial screening phase consisted of initial medical/dental and eligibility screening. Subjects then underwent an Oxygen Desaturation Index (ODI) screening (confirming ODI of 10-60) and one night of home use with the study device to screen for proper fit.
Groups:
- Sleep Apnea Treatment (Primary Endpoint Cohort): The Treatment group (Primary Endpoint Cohort) includes subjects with an evaluable control (without Attune system) and treatment (with Attune system) polysomnogram (PSG).
Period: Screening Cohort
Arm/Group | Sleep Apnea Treatment (Primary Endpoint Cohort)
Started | 367
Completed | 146
Not Completed | 221
Not completed — Screen Failure | 187
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 29
Period: Safety Cohort
Arm/Group | Sleep Apnea Treatment (Primary Endpoint Cohort)
Started | 146
Completed | 63
Not Completed | 83
Not completed — Screen Failure | 61
Not completed — Withdrawal by Subject | 4
Not completed — Control AHI <5 | 4
Not completed — TST <4 hrs | 14
Period: Primary Endpoint Cohort
Arm/Group | Sleep Apnea Treatment (Primary Endpoint Cohort)
Started | 63 (63 Subjects in the Primary Endpoint Cohort)
Completed | 57 (57 Subjects in the Primary Endpoint Cohort completed the 28 day study)
Not Completed | 6
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Baseline Demographics and Characteristics are presented for the Safety Cohort
Groups:
- Safety Cohort: Demographics and Baseline Characteristics are presented for the Safety Cohort (N=146)
Arm/Group | Safety Cohort
Number analyzed (Participants) | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 130
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 100
Region of Enrollment [Number; unit: participants]
  United States | 146

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success Defined as Apnea-hypopnea Index (AHI) Reduction of >50% and Treated AHI<20
Description: Comparing first treatment night AHI to control/baseline night. AHI is calculated by dividing the number of apnea/hypopnea events by the number of hours of sleep. AHI values are typically characterized as 5-15/hr = mild OSA, 15-30/hr = moderate OSA, and >30/hr = severe OSA. For each subject, Clinical success was defined as apnea-hypopnea index (AHI) reduction of >50% and treated AHI<20. The number of subjects with clinical success was determined to calculate the primary endpoint as the ratio of the number of subjects with clinical success to the number of subjects.
Time Frame: first treatment night
Population: All subjects in the primary endpoint cohort were analyzed.
Measure: Number; unit: subjects with clinical success
Groups:
- Primary Endpoint Cohort: The Treatment group (Primary Endpoint Cohort) includes subjects with an evaluable control (without Attune system) and treatment (with Attune system) PSG.
Arm/Group | Primary Endpoint Cohort
Number analyzed (Participants) | 63
subjects with clinical success | 26

2. Secondary Outcome: Adverse Event Rate
Description: Further categorized as serious and non-serious, device-related and non-device-related, unanticipated and anticipated, and based on level of severity. Adverse events will be evaluated during the trial at the following visits during 28-day take-home period: 7-day, 14-day, 21-day, 28-day follow-up, and any unscheduled visits.
Time Frame: 4 weeks
Population: The Safety Cohort consisted of all subjects who participated in at-home use of the device.
Measure: Number; unit: subjects
Groups:
- Safety Cohort: The Safety Cohort is comprised of all subjects with at least one night of Winx therapy usage.
Arm/Group | Safety Cohort
Number analyzed (Participants) | 146
subjects
  Unanticipated Adverse Events | 0
  All adverse events | 87
  Device related adverse events | 80
  Device related AEs categorized as mild | 65
  Device related AEs categorized as moderate | 15
  Device related AEs categorized as severe | 0
  Serious adverse events | 0

3. Secondary Outcome: Last Treatment Night Response (AHI Reduction)
Description: Comparing AHI at the last treatment night to the control/baseline night is reported as the percent change in AHI. AHI is calculated by dividing the number of apnea/hypopnea events by the number of hours of sleep. AHI values are typically characterized as 5-15/hr = mild OSA, 15-30/hr = moderate OSA, and >30/hr = severe OSA. Negative numbers represent a decrease/improvement in AHI, whereas positive numbers represent an increase/no improvement in AHI.
Time Frame: At completion of 28 day home use.
Population: All subjects in primary endpoint cohort with final evaluable treatment PSG.
Measure: Median (Inter-Quartile Range); unit: AHI reduction (% change)
Arm/Group | Primary Endpoint Cohort
Number analyzed (Participants) | 52
AHI reduction (% change) | -43.2 [-71.7 to 15.9]

4. Secondary Outcome: Percent Reduction in Oxygen Desaturation Index (ODI)
Description: Comparing first treatment night to control/baseline night reported as percent change. Negative numbers represent a reduction/improvement in ODI, whereas positive numbers represent increases/no improvement in ODI.
Time Frame: First treatment night
Measure: Median (Inter-Quartile Range); unit: ODI reduction (% change)
Arm/Group | Primary Endpoint Cohort
Number analyzed (Participants) | 63
ODI reduction (% change) | -41.9 [-63.5 to 9.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collect at screening, control and treatment PSG, 7 days, 14 days, 21 days, 28 days and after the final treatment PSG.
Groups:
- Safety Cohort: Device related adverse events are presented for the Safety Cohort.
Arm/Group | Safety Cohort
Serious Adverse Events (participants affected / at risk) | 0/146
Other Adverse Events (participants affected / at risk) | 80/146
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Cohort (N=146)
Oral Tissue Discomfort (Skin and subcutaneous tissue disorders) | 70
Oral Tissue Irritation (Skin and subcutaneous tissue disorders) | 27
Occlusal Change (General disorders) | 1
Dental Discomfort (General disorders) | 19
Excessive Salivation (General disorders) | 3
Other Adverse Event (General disorders) | 21 — Other AEs included: blood in mucous/saliva, headache, jaw discomfort, keratosis on tongue, leukoplakia, metallic taste in mouth, nasal congestion, nausea, panic attack.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No